CLINICAL TRIAL: NCT04062474
Title: Treatment of Pain in Patients With Lumbar Spinal Stenosis By Epidural Intervention of Spinal Nerves With Local Anesthetic, Steroids and Tumor Necrosis Factor-Alpha Inhibitor Respectively：a Prospective Randomized Study
Brief Title: Epidural Intervention of Spinal Nerves With Tumor Necrosis Factor-Alpha Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20151014-01
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-05

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural Intervention with Steroids (Experimental): Epidural Intervention with Steroids
  Interventions: Procedure: Epidural Intervention with TNF-α inhibitor

INTERVENTIONS:
Procedure: Epidural Intervention with TNF-α inhibitor — Epidural administration with TNF-α inhibitor

SUMMARY:
This study is to assess the clinical efficacy of epidural injections with Tumor Necrosis Factor-Alpha(TNF-α) Inhibitor in patients with chronic radicular pain caused by lumbar spinal stenosis.

DETAILED DESCRIPTION:
This study is to assess the clinical efficacy of epidural injections with Tumor Necrosis Factor-Alpha(TNF-α) Inhibitor in patients with chronic radicular pain caused by lumbar spinal stenosis.Ninety patients were diagnosed with lumbar spinal stenosis and were randomly assigned to 3 groups, for each group 30 cases. Patients in Group A received epidural injection of spinal nerve with 2.0 ml of lidocaine and 10 mg of Tumor Necrosis Factor-Alpha Inhibitor (etanercept) onto the affected spinal nerve, Group B patients received epidural injection with lidocaine 2ml mixed with 2ml of steroid(Diprospan), and group C patients received epidural injections with 4.0 ml of lidocaine only. All the 3 groups were evaluated by VAS and ODI, and received 6 months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinal stenosis with radicular pain at least 5 scores of VAS(ranging from 0 to 10).
* Failed to improve symptom significantly through conservative treatment, including physiotherapy, chiropractic therapy, exercise, medication and bed rest.

Exclusion Criteria:

* lumbar surgery history,
* spinal stenosis without radicular pain,
* uncontrollable or unstable use of opioids,
* uncontrolled mental illness,
* pregnant or lactating women,
* patients with a history of adverse reactions or possible adverse reactions to local anesthetics, etanercept or Steroids.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 6 months
  visual analog scale(0-10 scores) is for pain, 0 represent no pain, 10 score represent the severe pain.
Oswestry Disability Index | 6 months
  Oswestry Disability Index is for movement function, Questionnaire examines

REFERENCES:
- [Derived] Wei P, Xu Y, Yao Q, Wang L. Randomized trial of 3-drug combination for lumbar nerve root epidural injections with a TNF-alpha inhibitor in treatment of lumbar stenosis. Br J Neurosurg. 2020 Apr;34(2):168-171. doi: 10.1080/02688697.2020.1713990. Epub 2020 Jan 20. PMID 31955619